CLINICAL TRIAL: NCT00180700
Title: The Effects of Two Psychological Intervention Techniques, Self-hypnosis and Johrei Healing Method, on Quality of Life, Psychological Well-being, EEG Measures and Various Immunological Measures Including CD4+ Counts in Early HIV: a Randomly Controlled Pilot Study
Brief Title: The Influence of Psychological Interventions Upon Disease Progression in HIV-infected Patients Receiving no Medication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Hammersmith Hospitals NHS Trust (Other); Johrei Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Johrei_HIV1
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: HIV Infected Individuals
Keywords: HIV; Stress; Psychoneuroimmunology; stress management; hypnosis; Johrei; psychological intervention
MeSH Terms: interventions — Hypnosis

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-hypnosis (Experimental): A course of four weekly 2-hour training sessions coupled with daily self-hypnosis practice was given to 13 participants with diagnosed HIV
  Interventions: Behavioral: Hypnosis
- Johrei healing method (Experimental): A course of four weekly 2-hour training sessions coupled with daily self-hypnosis practice was given to 9 participants with diagnosed HIV
  Interventions: Behavioral: Hypnosis

INTERVENTIONS:
Behavioral: Hypnosis

SUMMARY:
This study examines the hypothesis that psychological interventions have beneficial effects on quality of life including psychological well-being and disease progression in early HIV patients recieving no medication.

DETAILED DESCRIPTION:
Hypothesis: This investigation is based upon the hypothesis that psychological intervention may counteract the detrimental effects of stress both on psychological well-being and on general health.

Background: HIV infection may be considered to be a life-long biological and psychological stressor leading to detrimental outcomes associated with disease progression. Stress reduction in these patients may have beneficial effects through delaying disease progression via the proposed interactive psycho-neuro-endocrine-immune network.

Inclusion Criteria:

HIV infected individuals CD4 T-cell counts above 200 cells/mcl Receiving no anti-retroviral drugs Individuals who signed the informed consent form

Investigative approach: Self-hypnosis and a Japanese non-touching, laying-on-of hands-like technique, called Johrei, were used to investigate the effects of psychological intervention upon immune parameters (especially in CD4 counts) associated with disease progression along with phenomenological associations between stress perception and stress hormone levels in HIV-infected patients receiving no medication.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* CD4 T-cell counts above 200 cells/mcl
* Signed the informed consent form

Exclusion Criteria:

* receiving anti-retroviral drugs

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2003-06-01 (Actual); Primary Completion 2003-12-01 (Actual); Study Completion 2003-12-01 (Actual)

PRIMARY OUTCOMES:
CD4 T-cell counts | 4 weeks
  Lab test

SECONDARY OUTCOMES:
Other immunological parameters (Viral load levels, NK cell counts) | 4 weeks
Psychological questionnaires (Perceived Stress Scale (PSS), STAI, Beck depression Inventory (BDI)) | 4 weeks
Endogenous hormone levels (cortisol, DHEA-S and melatonin) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John H Gruzelier, Ph.D., Principal Investigator — Imperial College London; Don C Henderson, Ph.D., Study Director — Imperial College London
Locations (1):
- Imperial College London, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No